CLINICAL TRIAL: NCT05192538
Title: A Novel Endoloop Pre-test to Treat Gastroesophageal Reflux Before Anti-reflux Surgery or Endoscopic Treatment
Brief Title: A Novel Endoloop Pre-test to Treat Gastroesophageal Reflux
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Beijing 302 Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE-Endoloop
Record Dates: First submitted 2021-11-29; First posted 2022-01-14 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: GERD; Reflux Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis, Peptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic endoloop pre-test treatment (Experimental): Endoscopic endoloop pre-test treatment is a less invasive reversible endoscopic treatment to predict whether the gastroesophageal reflux can be alleviated in order to ultimately decide whether to undergo irreversible surgery or endoscopic treatment.
  Interventions: Device: Endoscopic endoloop pre-test treatment

INTERVENTIONS:
Device: Endoscopic endoloop pre-test treatment — A novel endoloop was inserted into the gastric cardia by forceps through the single-channel endoscopy. After adjustment of the endoloop's location and angle, it was anchored onto the edge of the gastric cardia with clip and another 1 or 2 clips were inserted to hold the opposite side of endoloop at about 1/2 circumference. Then the hook was connected with the endoloop, which was tighted by slight pulling together of all the clips.

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of endoscopic endoloop pre-test for gastroesophageal reflux before anti-reflux surgery or endoscopic treatment. In the study, the investigators used the novel pre-test to narrow the gastric cardia to control symptoms temporarily to decide whether to undergo irreversible surgery or endoscopic treatment.Thirty patients were enrolled and underwent endoscopic endoloop pre-test treatment. The Primary outcome in this study was measured by the percent reduction in post-procedure GERD symptoms as evidenced by analysis of the GERD-HRQL (Health Related Quality of Life) questionnaire. The secondary outcomes included improvement in esophageal 24-hr pH monitoring, improvement in quality of life questionnaires and safety. Patient follow-up assessments were completed at 7 and 14 days post treatment.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a neuromuscular disorder with abnormal reflux of gastric contents into the esophagus.The most common symptoms are heartburn, dysphagia, and regurgitation.Due to less invasion, several endoscopic treatments of GERD have been investigated, such as collagen or radio frequency delivery, and antireflux mucosectomy(ARMS).The disadvantages of these treatment included short-term effectiveness, increasing reflux and ulcer, and serious complications. A novel endoscopic endoloop pre-test treatment has been developed, offering a minimally reversible endoscopic treatment to predict whether the symptoms can be alleviated in order to ultimately decide whether to undergo irreversible surgery or endoscopic treatment, which can be performed in an outpatient setting.The aim of this study was to assess the feasibility and safety of the pre-test treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with typical symptoms of GERD with symptomatic response to PPI therapy for ≥ 3 months
* Patients considered for non-medical therapy, i.e. unwillingness to take life-long medication in medically-responding disease, suffering from medication side-effects or medically-intractable disease
* Pathological esophageal acid exposure after discontinuation of medical therapy, proven by ambulatory 24-hour pH-monitoring with > 5% of time a pH < 4 and a symptom-association probability > 95%
* written informed consent

Exclusion Criteria:

* 24 hr acid exposure study showing abnormal esophageal acid exposure <4%
* DeMeester Score <14.7
* hiatal hernia (> 3 cm in length)
* history of antireflux or esophageal/gastric surgery
* severe psychiatric disease
* Barrett's esophagus with dysplasia
* esophageal stenosis/malignancy
* pregnancy or lactation
* history of low therapeutic compliance
* other severe comorbidity (including cardiopulmonary disease, portal hypertension, collagen diseases, morbid obesity, coagulation disorder)
* use of anticoagulant or immunosuppressive drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in GERD-Health Related Quality of Life (HRQL) questionnaire scores | 3 days
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
Improvement in GERD-Health Related Quality of Life (HRQL) questionnaire scores | 7 days
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
Improvement in GERD-Health Related Quality of Life (HRQL) questionnaire scores | 14 days
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
Improvement in GERD-Health Related Quality of Life (HRQL) questionnaire scores | 21 days
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
Improvement in GERD-Health Related Quality of Life (HRQL) questionnaire scores | 1 month
  GERD-HRQL is a validate questionnaire to evaluate GERD-related esophageal symptoms. The scale range is (0-50); the higher values represents worse outcomes.
Improvement in Reflux Symptom Index (RSI) questionnaire scores | 3 days
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
Improvement in Reflux Symptom Index (RSI) questionnaire scores | 7 days
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
Improvement in Reflux Symptom Index (RSI) questionnaire scores | 14 days
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
Improvement in Reflux Symptom Index (RSI) questionnaire scores | 21 days
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.
Improvement in Reflux Symptom Index (RSI) questionnaire scores | 1 month
  RSI is a validate questionnaire to evaluate GERD-related extra- esophageal symptoms. The scale range is (0-45); the higher values represents worse outcomes.

SECONDARY OUTCOMES:
Effect on 24-hours esophageal pH-impedance | 7 days
  Parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
Effect on 24-hours esophageal pH-impedance | 14 days
  Parameter detected by 24hours esophagel pH-metry. pH-metric and impedance parameters are indicators of procedure effectiveness as able to quantify the presence of gastro-esophageal reflux.
Changes in DeMeester score | 7 days
  DeMeester score is a composite score which examined six variables (number of reflux episodes, number of episodes longer than 5 minutes, longest reflux duration, total percentage of monitoring time with pH below 4, and the percentage of time with pH below 4 in an upright position and supine position). A score of >14.72 shows a pathological reflux. Higher values represent worse outcomes.
Changes in DeMeester score | 14 days
  DeMeester score is a composite score which examined six variables (number of reflux episodes, number of episodes longer than 5 minutes, longest reflux duration, total percentage of monitoring time with pH below 4, and the percentage of time with pH below 4 in an upright position and supine position). A score of >14.72 shows a pathological reflux. Higher values represent worse outcomes.
Safety and Tolerability of the procedure | 7 days
  Incidence of Treatment-Emergent Adverse Events
Safety and Tolerability of the procedure | 14 days
  Incidence of Treatment-Emergent Adverse Events
Safety and Tolerability of the procedure | 1 month
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Pro., Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No